CLINICAL TRIAL: NCT00005500
Title: Collaborative Studies on the Genetics of Asthma (CSGA)
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 5018; U01HL049609 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
To conduct molecular genetic studies in human pedigrees in order to identify the major genes responsible for asthma.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a respiratory disease characterized by variable airways obstruction, airways inflammation and bronchial hyperresponsiveness (BHR). There are recent increases in asthma mortality and prevalence in the US, especially in African-Americans. Multiple studies suggest that both genetic and environmental factors are important in asthma susceptibility.

The study was recommended by the Pulmonary Diseases Advisory Committee at its February 1991 meeting and given concept approval by the May 1991 National Heart, Lung, and Blood Advisory Council. The Request for Applications was released in October 1992.

DESIGN NARRATIVE:

The CSGA was composed of five centers (Johns Hopkins University, University of Chicago, University of Maryland, University of Minnesota, and a data coordinating center at Wake Forest). At each center, families were ascertained through two siblings with asthma. All family members were characterized with spirometry, bronchial responsiveness to methacholine or reversibility testing, skin-tests and questionnaire data. The initial genome screen was completed on the first 237 sib pairs from three racial groups (African-American, Caucasian and Hispanic), and genotyping on the remaining family members and families was completed before the study was renewed in 1997. Therefore, the initial aim of the CSGA to map susceptibility regions was completed, with detection of several novel chromosomal regions, and replication of several regions previously linked to associated phenotypes.

In order to determine the importance of these regions in asthma susceptibility and the impact of environmental rink factors, the investigators l) evaluated the evidence for linkage in the complete CSGA data using 2-point, multipoint and multilocus approaches for asthma and associated phenotypes (including BHR, total serum IgE and skin test reactivity to standardized allergens); 2) performed fine mapping studies of regions using additional genetic markers to obtain a < 2 cM map; 3) identified candidate genes and novel sequence variants; and 4) characterized a patient population with asthma to study identified variants with respect to asthma severity and bronchial inflammation. These studies allowed identification of asthma susceptibility genes and their variants, interactions with other genes and environmental risk factors, as well as provided insight for the development of improved treatment and ultimate prevention of asthma.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1992-09; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri Beatty — Johns Hopkins University; Eugene Bleecker — University of Maryland; Malcolm Blumenthal — University of Minnesota; Carole Ober — University of Chicago; Stephen Rich — Wake Forest University

REFERENCES:
- [Background] Bleecker ER, Postma DS, Meyers DA. Genetic susceptibility to asthma in a changing environment. Ciba Found Symp. 1997;206:90-9; discussion 99-105, 106-10. doi: 10.1002/9780470515334.ch6. PMID 9257007
- [Background] A genome-wide search for asthma susceptibility loci in ethnically diverse populations. Nat Genet. 1997 Apr;15(4):389-92. doi: 10.1038/ng0497-389. PMID 9090385
- [Background] Marsh DG. Approaches toward the genetic analysis of complex traits: asthma and atopy. Am J Respir Crit Care Med. 1997 Oct;156(4 Pt 2):S133-8. doi: 10.1164/ajrccm.156.4.12tac11. PMID 9351594
- [Background] Blumenthal MN, Rich SS, King R, Weber J. Approaches and issues in defining asthma and associated phenotypes map to chromosome susceptibility areas in large Minnesota families. The Collaborative Study for the Genetics of Asthma (CSGA). Clin Exp Allergy. 1998 Apr;28 Suppl 1:51-5; discussion 65-6. doi: 10.1046/j.1365-2222.1998.0280s1051.x. PMID 9641593
- [Background] Hizawa N, Collins G, Rafnar T, Huang SK, Duffy DL, Weber JL, Freidhoff LR, Ehrlich E, Marsh DG, Beaty TH, Barnes KC. Linkage analysis of Dermatophagoides pteronyssinus-specific IgE responsiveness with polymorphic markers on chromosome 6p21 (HLA-D region) in Caucasian families by the transmission/disequilibrium test. Collaborative Study on the Genetics of Asthma (CSGA). J Allergy Clin Immunol. 1998 Sep;102(3):443-8. doi: 10.1016/s0091-6749(98)70133-2. PMID 9768586
- [Background] Ober C, Cox NJ, Abney M, Di Rienzo A, Lander ES, Changyaleket B, Gidley H, Kurtz B, Lee J, Nance M, Pettersson A, Prescott J, Richardson A, Schlenker E, Summerhill E, Willadsen S, Parry R. Genome-wide search for asthma susceptibility loci in a founder population. The Collaborative Study on the Genetics of Asthma. Hum Mol Genet. 1998 Sep;7(9):1393-8. doi: 10.1093/hmg/7.9.1393. PMID 9700192
- [Background] Mathias RA, Freidhoff LR, Blumenthal MN, Meyers DA, Lester L, King R, Xu JF, Solway J, Barnes KC, Pierce J, Stine OC, Togias A, Oetting W, Marshik PL, Hetmanski JB, Huang SK, Ehrlich E, Dunston GM, Malveaux F, Banks-Schlegel S, Cox NJ, Bleecker E, Ober C, Beaty TH, Rich SS; CSGA (Collaborative Study of the Genetics of Asthma). Genome-wide linkage analyses of total serum IgE using variance components analysis in asthmatic families. Genet Epidemiol. 2001 Apr;20(3):340-55. doi: 10.1002/gepi.5. PMID 11255243
- [Background] Barnes KC, Freidhoff LR, Horowitz EM, Mathias RA, Mulkern DM, Bonacum JT, Goldman MH, Polito AJ, Saini SS, Marsh DG, Beaty TH, Togias A. Physician-derived asthma diagnoses made on the basis of questionnaire data are in good agreement with interview-based diagnoses and are not affected by objective tests. J Allergy Clin Immunol. 1999 Oct;104(4 Pt 1):791-6. doi: 10.1016/s0091-6749(99)70289-7. PMID 10518823
- [Background] Xu J, Meyers DA, Ober C, Blumenthal MN, Mellen B, Barnes KC, King RA, Lester LA, Howard TD, Solway J, Langefeld CD, Beaty TH, Rich SS, Bleecker ER, Cox NJ; Collaborative Study on the Genetics of Asthma. Genomewide screen and identification of gene-gene interactions for asthma-susceptibility loci in three U.S. populations: collaborative study on the genetics of asthma. Am J Hum Genet. 2001 Jun;68(6):1437-46. doi: 10.1086/320589. Epub 2001 May 10. PMID 11349227
- [Background] Langefeld CD, Davis CC, Brown WM. Nonparametric linkage regression. I: Combined Caucasian CSGA and German genome scans for asthma. Genet Epidemiol. 2001;21 Suppl 1:S136-41. doi: 10.1002/gepi.2001.21.s1.s136. PMID 11793656
- [Background] Davis CC, Brown WM, Lange EM, Rich SS, Langefeld CD. Nonparametric linkage regression. II: Identification of influential pedigrees in tests for linkage. Genet Epidemiol. 2001;21 Suppl 1:S123-9. doi: 10.1002/gepi.2001.21.s1.s123. PMID 11793654
- [Background] Meyers DA, Wjst M, Ober C. Description of three data sets: Collaborative Study on the Genetics of Asthma (CSGA), the German Affected-Sib-Pair Study, and the Hutterites of South Dakota. Genet Epidemiol. 2001;21 Suppl 1:S4-8. doi: 10.1002/gepi.2001.21.s1.s4. PMID 11793707
- [Background] Marsh DG. Approaches toward the genetic analysis of complex traits: asthma and atopy. Allergy. 1999 Mar;54(3):198-205. doi: 10.1034/j.1398-9995.1999.00090.x. PMID 10321554
- [Background] Nickel RG, Saitta FP, Freidhoff LR, Yu XY, Ehrlich E, Barnes KC, Beaty T, Huang SK. Positional candidate gene approach and functional genomics strategy in atopy gene discovery. Int Arch Allergy Immunol. 1999 Feb-Apr;118(2-4):282-4. doi: 10.1159/000024100. PMID 10224411
- [Background] Ober C, Leavitt SA, Tsalenko A, Howard TD, Hoki DM, Daniel R, Newman DL, Wu X, Parry R, Lester LA, Solway J, Blumenthal M, King RA, Xu J, Meyers DA, Bleecker ER, Cox NJ. Variation in the interleukin 4-receptor alpha gene confers susceptibility to asthma and atopy in ethnically diverse populations. Am J Hum Genet. 2000 Feb;66(2):517-26. doi: 10.1086/302781. PMID 10677312
- [Background] Howard TD, Meyers DA, Bleecker ER. Mapping susceptibility genes for asthma and allergy. J Allergy Clin Immunol. 2000 Feb;105(2 Pt 2):S477-81. doi: 10.1016/s0091-6749(00)90046-0. PMID 10669527
- [Background] Howard TD, Bleecker ER, Stine OC. Fluorescent allele-specific PCR (FAS-PCR) improves the reliability of single nucleotide polymorphism screening. Biotechniques. 1999 Mar;26(3):380-1. doi: 10.2144/99263bm01. No abstract available. PMID 10090967
- [Background] Stine OC, Xu J, Meyers DA, Bleecker ER. Approaches to fine mapping in asthma. Clin Exp Allergy. 1998 Apr;28 Suppl 1:98-100; discussion 108-10. doi: 10.1046/j.1365-2222.1998.0280s1098.x. No abstract available. PMID 9641604
- [Background] Ober C. Susceptibility genes in asthma and allergy. Curr Allergy Asthma Rep. 2001 Mar;1(2):174-9. doi: 10.1007/s11882-001-0085-4. PMID 11899300
- [Background] Ober C, Abney M, McPeek MS. The genetic dissection of complex traits in a founder population. Am J Hum Genet. 2001 Nov;69(5):1068-79. doi: 10.1086/324025. Epub 2001 Oct 3. PMID 11590547
- [Background] Wu X, Di Rienzo A, Ober C. A population genetics study of single nucleotide polymorphisms in the interleukin 4 receptor alpha (IL4RA) gene. Genes Immun. 2001 May;2(3):128-34. doi: 10.1038/sj.gene.6363746. PMID 11426321
- [Background] Abney M, McPeek MS, Ober C. Broad and narrow heritabilities of quantitative traits in a founder population. Am J Hum Genet. 2001 May;68(5):1302-7. doi: 10.1086/320112. Epub 2001 Apr 10. PMID 11309690
- [Background] Ober C, Tsalenko A, Parry R, Cox NJ. A second-generation genomewide screen for asthma-susceptibility alleles in a founder population. Am J Hum Genet. 2000 Nov;67(5):1154-62. doi: 10.1016/S0002-9297(07)62946-2. Epub 2000 Oct 5. PMID 11022011
- [Background] Summerhill E, Leavitt SA, Gidley H, Parry R, Solway J, Ober C. beta(2)-adrenergic receptor Arg16/Arg16 genotype is associated with reduced lung function, but not with asthma, in the Hutterites. Am J Respir Crit Care Med. 2000 Aug;162(2 Pt 1):599-602. doi: 10.1164/ajrccm.162.2.9910108. PMID 10934093
- [Background] Donfack J, Tsalenko A, Hoki DM, Parry R, Solway J, Lester LA, Ober C. HLA-DRB1*01 alleles are associated with sensitization to cockroach allergens. J Allergy Clin Immunol. 2000 May;105(5):960-6. doi: 10.1067/mai.2000.106926. PMID 10808177
- [Background] Abney M, McPeek MS, Ober C. Estimation of variance components of quantitative traits in inbred populations. Am J Hum Genet. 2000 Feb;66(2):629-50. doi: 10.1086/302759. PMID 10677322
- [Background] Ober C, Tsalenko A, Willadsen S, Newman D, Daniel R, Wu X, Andal J, Hoki D, Schneider D, True K, Schou C, Parry R, Cox N. Genome-wide screen for atopy susceptibility alleles in the Hutterites. Clin Exp Allergy. 1999 Dec;29 Suppl 4:11-5. PMID 10641559
- [Background] Blumenthal MM. What we know about the genetics of asthma at the beginning of the 21st century. Clin Rev Allergy Immunol. 2002 Feb;22(1):11-31. doi: 10.1007/s12016-002-0003-0. PMID 11803799
- [Background] Donfack J, Kogut P, Forsythe S, Solway J, Ober C. Sequence variation in the promoter region of the cholinergic receptor muscarinic 3 gene and asthma and atopy. J Allergy Clin Immunol. 2003 Mar;111(3):527-32. doi: 10.1067/mai.2003.71. PMID 12642833
- [Background] Huang SK, Mathias RA, Ehrlich E, Plunkett B, Liu X, Cutting GR, Wang XJ, Li XD, Togias A, Barnes KC, Malveaux F, Rich S, Mellen B, Lange E, Beaty TH; Comparative Study on the Genetics of Asthma. Evidence for asthma susceptibility genes on chromosome 11 in an African-American population. Hum Genet. 2003 Jul;113(1):71-5. doi: 10.1007/s00439-003-0934-4. Epub 2003 Mar 27. PMID 12664305
- [Background] Hsu FC, Liang KY, Beaty TH. Multipoint linkage disequilibrium mapping approach: incorporating evidence of linkage and linkage disequilibrium from unlinked region. Genet Epidemiol. 2003 Jul;25(1):1-13. doi: 10.1002/gepi.10241. PMID 12813722
- [Background] Colilla S, Nicolae D, Pluzhnikov A, Blumenthal MN, Beaty TH, Bleecker ER, Lange EM, Rich SS, Meyers DA, Ober C, Cox NJ; Collaborative Study for the Genetics of Asthma. Evidence for gene-environment interactions in a linkage study of asthma and smoking exposure. J Allergy Clin Immunol. 2003 Apr;111(4):840-6. doi: 10.1067/mai.2003.170. PMID 12704367
- [Background] Blumenthal MN, Langefeld CD, Beaty TH, Bleecker ER, Ober C, Lester L, Lange E, Barnes KC, Wolf R, King RA, Solway J, Oetting W, Meyers DA, Rich SS. A genome-wide search for allergic response (atopy) genes in three ethnic groups: Collaborative Study on the Genetics of Asthma. Hum Genet. 2004 Jan;114(2):157-64. doi: 10.1007/s00439-003-1030-5. Epub 2003 Oct 25. PMID 14586638
- [Background] Lester LA, Rich SS, Blumenthal MN, Togias A, Murphy S, Malveaux F, Miller ME, Dunston GM, Solway J, Wolf RL, Samet JM, Marsh DG, Meyers DA, Ober C, Bleecker ER; Collaborative Study on the Genetics of Asthma. Ethnic differences in asthma and associated phenotypes: collaborative study on the genetics of asthma. J Allergy Clin Immunol. 2001 Sep;108(3):357-62. doi: 10.1067/mai.2001.117796. PMID 11544453
- [Background] Liang KY, Hsu FC, Beaty TH. Multipoint linkage disequilibrium mapping for complex diseases. Genet Epidemiol. 2003 Dec;25(4):285-92. doi: 10.1002/gepi.10271. PMID 14639698
- [Background] Blumenthal MN, Ober C, Beaty TH, Bleecker ER, Langefeld CD, King RA, Lester L, Cox N, Barnes K, Togias A, Mathias R, Meyers DA, Oetting W, Rich SS; CSGA. Genome scan for loci linked to mite sensitivity: the Collaborative Study on the Genetics of Asthma (CSGA). Genes Immun. 2004 May;5(3):226-31. doi: 10.1038/sj.gene.6364063. PMID 15029235
- [Background] Blumenthal MN, Langefeld CD, Barnes KC, Ober C, Meyers DA, King RA, Beaty TH, Beck SR, Bleecker ER, Rich SS; Collaborative Study on the Genetics of Asthma. A genome-wide search for quantitative trait loci contributing to variation in seasonal pollen reactivity. J Allergy Clin Immunol. 2006 Jan;117(1):79-85. doi: 10.1016/j.jaci.2005.09.038. PMID 16387588